CLINICAL TRIAL: NCT06057961
Title: The Effect of Art Therapy Applied to Individuals With Substance Use Subject To Supervised Release on Emotion Regulation Difficulties, Self-Esteem and Hopeless
Brief Title: Effect Of Art Therapy Applied to Individuals With Substance Use Subject to Supervised Release
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Seval Cüceler, MSc, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MersinU-SC-01
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Substance Use
Keywords: Substance Use; Probation; Art therapy; Psychiatric Nursing
MeSH Terms: conditions — Substance-Related Disorders | interventions — Art Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): "Personal Information Form", "Difficulties in Emotion Regulation Scale-Brief Form (DERS-16)", "Coopersmith Self-Esteem Scale", "Beck Hopelessness Scale" will be applied to the intervention group as part of the pre-test application. In the research, art therapy will be applied face to face to the participants in the intervention group, in groups of 4-12 people, in the group guide room, on a common day and time determined by the group members and the researchers.The art therapy to be applied to the participants in the intervention group in the study consists of eight sessions.Each session is planned to last approximately 60-90 minutes.
  Interventions: Other: Art Therapy
- Control (No Intervention): Individuals who meet the inclusion criteria and agree to participate in the research will be informed about the research and their verbal and written consent will be obtained. Interviews will be held to implement the pre-tests ("Personal Information Form", "Emotion Regulation Difficulties Scale-Short Form (DERS-16)", "Coopersmith Self-Esteem Scale", "Beck Hopelessness Scale"). A session will be held to implement the post-tests and to implement the "Awareness of Emotions" themed session with the intervention group to the control group.

INTERVENTIONS:
Other: Art Therapy — 8 meetings in 1 year
  Arms: Experimental

SUMMARY:
The goal of this clinical trial is to examine the effect of art therapy applied to individuals with substance use who are subject to probation on difficulty in emotion regulation, self-esteem and hopelessness. The main question[s] it aims to answer are:

[Is art therapy effective on the level of emotion regulation difficulties of individuals with substance use who are subject to probation?] [Is art therapy effective on the self-esteem level of individuals with substance use who are subject to probation?][Is art therapy effective on the hopelessness level of individuals with substance use who are subject to probation?] Data will be collected through scale forms and art therapy sessions. Within the scope of the pre-test application, data will be collected from all participants in the sample group using the "Personal Information Form", "Difficulties in Emotion Regulation Scale-Brief Form (DERS-16)", "Coopersmith Self-Esteem Scale", "Beck Hopelessness Scale". Art therapy will be applied face to face to the participants in the intervention group, in groups of 4-12 people, in the group guide room, on a common day and time determined by the group members and the researchers.

Researchers will compare the experimental group and the control group to see whether art therapy applied to individuals with substance use who are subject to probation has an effect on emotion regulation difficulties, self-esteem and hopelessness.

DETAILED DESCRIPTION:
Substance use is an important public health problem that negatively affects the health of the individual and the environment, has criminal, economic and social dimensions and is increasingly prevalent all over the world .According to the 2022 world drug report of the United Nations Office on Drugs and Crime; In 2020, an estimated 284 million individuals aged 15-64 years (mostly men) worldwide have used drugs in the past 12 months .In addition, according to the 2022 Turkey drug report, there are 100,140 convicts and detainees in penal institutions due to drug-related crimes as of 2021 .According to the data of the Ministry of Justice, the number of individuals under Treatment and Probation due to crimes of using and possessing drugs and stimulants is reported to be 66,825 as of August 2022. Substance use has many negative effects on individuals. Substance use affects the central nervous system and organs, causes distortions in reality assessment, and causes physiological and psychological dependence over time. Individuals' education may be left unfinished, they may experience unemployment problems, and individuals may experience problems within the family (such as domestic violence, conflict between spouses). ) may encounter. Individuals may experience psychological problems such as loneliness, feeling of exclusion, anger, depression and anxiety, and may exhibit suicide, violence and criminal behavior. Additionally, individuals face legal sanctions due to illegal substance use. Another important problem experienced by individuals who use substances is difficulty in regulating emotions. Emotion regulation is defined by Gratz and Roomer (2004) as "the ability to be aware and understand emotions, accept emotions, control impulsive behaviors, and act in line with desired goals when experiencing negative emotions" and "to change emotional reactions as desired in order to meet individual goals and situational needs." It is explained as "the ability to flexibly use emotion regulation strategies appropriate to the situation". The absence of any or all of these skills indicates difficulty in regulating emotion. Individuals with emotion regulation difficulties have difficulty controlling their impulsive behavior in the face of negative emotions, maintaining their goal-oriented behavior, and accessing adaptive emotion regulation strategies .When emotion regulation difficulties are examined in terms of substance use; Individuals have difficulty in developing appropriate coping skills in the face of a negative emotion or situation and see substances as a coping method. They turn to substances to escape from the emotions they cannot regulate and, as a result, experience addiction-related problems. Addicted individuals experience many negative emotions such as shame, guilt, worthlessness and inadequacy.It is inevitable that individuals who have difficulty regulating these negative emotions use substances as a coping method. Difficulty in emotional regulation can negatively affect individuals who use substances in many ways. A study revealed that addicted individuals have difficulty controlling their impulses and acting goal-oriented while experiencing negative emotions, and this increases the severity of addiction .Another study reported that substance use increases impulsivity as well as difficulty in emotion regulation .Another study revealed a significant relationship between difficulty in emotion regulation and craving. In addition, individuals may experience stress-related impulse control problems related to difficulty in emotional regulation, which may lead to relapse. In addition to all these, there is a negative relationship between difficulty in emotion regulation and self-esteem .

Self-esteem is explained as an individual's general evaluation of his or her own worth. In general, they are positive or negative emotional states that an individual reaches as a result of self-evaluation. It is reported that self-esteem is low in individuals who use substances. A study reveals that self-esteem is low in individuals who apply to the probation unit due to substance use. Chronic substance use causes social relations to deteriorate, individuals to experience feelings of helplessness and inadequacy, and to isolate themselves from society and become lonely. Additionally, in a study, the rate of people who thought they were socially excluded due to substance use was found to be 84%. Individuals who are excluded from society and become lonely also have low self-esteem, which makes them even more lonely . It will be inevitable for an individual who becomes lonely and experiences conflicts in interpersonal relationships to turn to substances in order to cope with the social problems he experiences. In addition, low self-esteem can cause depression and anxiety in individuals. In a study, it was concluded that as self-esteem decreases, suicidal tendencies increase. It is also stated that low self-esteem leads individuals to crime and substance use. Individuals may tend to use substances to meet their self-esteem needs and to control their emotions and behaviors . In addition to all these, it has been reported that the level of hopelessness increases as the self-esteem of individuals using substances decreases.

Hope is seen as an effective coping mechanism that gives the individual strength to adapt to the future, increases his motivation, prevents feelings of pessimism and helplessness in case of illness, and increases compliance with treatment. Hopelessness is the feeling that the individual will not experience positive emotions or that there will be no improvement in his/her situation. Substance use and hopelessness mutually affect each other. In one study, individuals with high levels of hopelessness were found to be more likely to use substances at an early age, while in another study, it was found that the hopelessness level of individuals using substances was higher than those who did not use substances. Hopelessness negatively affects individuals in many ways. An individual who regrets substance use may feel hopeless, which pushes individuals to use substances again, causing a vicious circle. In addition, hopelessness can cause depression, and depression and substance use disorder can coexist. For this reason, addressing hopelessness in the treatment of individuals using substances is also important in preventing the development and progression of depression in individuals. In addition, hopelessness is seen as an important risk factor for completed suicide, suicide attempts and suicidal ideation, and it has been reported that suicidal thoughts increase as the hopelessness level of individuals using substances increases. As result, hopelessness negatively affects the quality of life of individuals who use substances.

In conclusion; Considering the devastating effects of difficulty in emotion regulation, low self-esteem, and hopelessness on individuals who use substances, it is of great importance that psychiatric nurses, who are important members of the mental health team, carry out intervention studies that address the difficulty in emotion regulation, self-esteem, and hopelessness of individuals who use substances. When the literature is examined, no intervention study based on art therapy has been found to date, in which three cases of individuals using substances are examined simultaneously. Therefore, in this study, art therapy, which reflects the inner world of individuals, provides the opportunity to regulate emotional experiences and expressions, mediates hope, causes a positive development in individuals and reduces physical and psychological problems, will be applied in a group environment to individuals with substance use who are subject to probation. Group counseling for individuals with substance use problems; This study will be conducted in a group environment, as it provides many benefits such as positive peer support, morale, reduced feeling of isolation, observation of improvement in peers and the creation of a sense of universality. In addition, art therapy; It helps individuals who use substances to overcome resistance, express difficult emotions, and develop a deep understanding of life. It is also stated that individuals with substance use who are subject to probation have difficulty in expressing themselves verbally and that art is an alternative way out in this regard. Art therapy offers individuals the opportunity to self-strengthen in a probation environment and opens a safe space to release their emotions. Considering all these, it is thought that it would be appropriate to apply art therapy to this sample group, and this study predicts that art therapy applied to individuals with substance use who are subject to probation will make positive contributions to the individuals' difficulty in emotion regulation, self-esteem and hopelessness.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are subject to probation within the scope of Article 191 of the Turkish Penal Code (purchasing, accepting or possessing drugs or stimulants for use, or using drugs or stimulants) between 2023-2024
* Literate
* Agreeing to participate in the research
* Those aged 18 and over
* Not under the influence of drugs
* In accordance with the Probation Services Regulation , individuals who are deemed ready for group work as a result of individual interviews conducted by the probation specialist.
* Individuals who do not have problems in terms of hearing, speaking and understanding that would prevent communication in the application to be performed.

Exclusion Criteria:

* Illiterate
* Under 18 years of age
* Under the influence of drugs
* In accordance with the Probation Services Regulation , individuals who are deemed not ready for group work as a result of individual interviews conducted by the probation specialist
* Individuals with hearing, speaking and understanding problems that will prevent communication in the application to be performed.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Difficulties in Emotion Regulation Scale-Brief Form (DERS-16) | Basseline and 8 weeks
  The Emotion Regulation Difficulty Scale-Short Form (DDGÖ-16), which is the short form of the Emotion Regulation Difficulty Scale developed by Gratz and Roemer (2004) to measure difficulties in regulating emotions, was developed by Bjureberg et al. (2016). The Turkish adaptation of DDGÖ-16 was made by Yiğit and Güzey Yiğit (2017). The Lilkert type scale consists of 16 items and is scored by grading the items between 1 (almost never) and 5 (almost always). There are no reverse coded items in the scale and there is no cut-off point. Scale, openness (1,2), goals (3,7,15), drive (4, 8,11), strategies (5, 6, 12, 14, 16), and nonacceptance (9, 10, 13). It consists of 5 sub-dimensions. High scores indicate greater difficulty in emotional regulation.
Coopersmith Self-Esteem Scale | Basseline and 8 weeks
  The scale was prepared by Stanley Copersmith in 1986 and was developed to be applicable to various age groups, especially adults. The reliability and validity study in our country was conducted by Tufan and Turan and the test-retest reliability of the scale was found to be 0.65 and 0.76. The scale consists of 25 items and the items are marked as "like me" or "not like me". The items include statements about the individual's perspective on life, family relationships, social relationships and endurance. The scores obtained vary between 0 and 100, and evaluation is made according to whether self-esteem is lower or higher than average. A score below the average indicates low self-esteem, while a score above the average indicates high self-esteem
Beck Hopelessness Scale | Basseline and 8 weeks
  Beck Hopelessness Scale, which measures the individual's negative expectations for the future, consists of a total of 20 items. The answer was "yes" to 11 of the items in the scale (Questions 2, 4, 7, 9, 11, 12, 14, 16, 17, 18, and 20), and to 9 items (Questions 1, 3, 5, 6, 8, (questions 10, 13, 15, and 19) are given one point each for a "no" answer. The lowest score to be obtained from the scale is 0 and the highest score is 20. High scores from the scale indicate that the individual's hopelessness is high.

CONTACTS AND LOCATIONS:
Overall Officials: Seval Cüceler, PhD, Principal Investigator — Toros University, Faculty of Health Sciences, Department of Nursing
Locations (1):
- Mersin Probation Directorate, Mersin, Akdeniz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.